CLINICAL TRIAL: NCT01094041
Title: Gluten Intolerance in Irritable Bowel Syndrome With Diarrhea: The Role of HLA-DQ2
Brief Title: Gluten Intolerance in Patients With Diarrhea Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-007344
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Diarrhea; Diarrhea Predominant Irritable Bowel Syndrome
Keywords: Gluten; Diarrhea or diarrhea predominant irritable bowel syndrome; Colonic permeability; Small bowel permeability; Colonic inflammatory response; Small bowel inflammatory response
MeSH Terms: conditions — Diarrhea | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten free diet (Experimental)
  Interventions: Other: Gluten free diet
- Gluten rich diet (Experimental)
  Interventions: Other: Gluten rich diet

INTERVENTIONS:
Other: Gluten free diet — A 4-week gluten free diet provided
  Arms: Gluten free diet
Other: Gluten rich diet — A 4-week gluten rich diet is provided
  Arms: Gluten rich diet

SUMMARY:
The specific hypotheses are:

Gluten supplementation for four weeks increases small intestinal permeability and accelerates colonic transit in patients with irritable bowel syndrome with diarrhea (IBS-D) or functional diarrhea (FD) who are HLA-DQ2 positive.

DETAILED DESCRIPTION:
The study design is a double-blind, randomized, controlled, parallel-group, 6-week study comparing the effects of gluten rich versus gluten free diets in diarrhea or diarrhea predominant IBS patients. All participants will keep a daily bowel pattern diary throughout the study. All participants will have negative serum tissue transglutaminase (TTg) assay, and anti-endomysial antibody test, if TTg is positive or equivocal. All participants will have the following studies performed both before and after the 4-week dietary intervention:

1. Stool samples to check markers of inflammation such as fecal calprotectin.
2. Blood samples to check markers of inflammation and for genetic testing.
3. After ingestion of the mannitol, lactulose and sucralose sugars, urine samples to indirectly measure small intestinal and colonic permeability.
4. After sedation, upper gastrointestinal endoscopy and flexible sigmoidoscopy to obtain 6 mucosal biopsies from the small bowel and sigmoid colon for immunohistochemical analysis.
5. Scintigraphy to measure gastrointestinal transit.

ELIGIBILITY:
Inclusion criteria:

1. Diarrhea or diarrhea predominant IBS patients
2. Age 18 to 65
3. BDQ confirms presence of IBS-D or functional diarrhea, positive by Rome III criteria
4. No restrictions on Hospital Anxiety Depression score
5. No abdominal surgery (except appendectomy and cholecystectomy)

Exclusion criteria:

1. Serum tissue transglutaminase IgA or IgG positive or medical record of small bowel biopsy suggestive of celiac disease
2. Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
3. Use of NSAIDs or aspirin within the past week (since NSAIDs affect intestinal permeability)
4. Use of oral corticosteroids within the previous 6 weeks
5. Ingestion of artificial sweeteners such as SplendaTM (sucralose), Nutrasweet TM(aspartame), lactulose or mannitol 2 days before the study begins, e.g., foods to be avoided are sugarless gums or mints and diet soda
6. Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before study begins.
7. Any females who are pregnant or trying to become pregnant (due to radiation exposure)
8. Bleeding disorders or medications that increase risk of bleeding from mucosal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Small bowel permeability | 0 - 2 hours post sugar ingestion
  Excretion of mannitol 0-2 hours after liquid formulation
Colonic permeability | 2 -24 hours post sugars ingestion
  Cumulative excretion of mannitol at 2-24 hours after liquid
Colonic transit | 24 hours
  Colonic transit geometric center at 24 hours

SECONDARY OUTCOMES:
Colon transit | 6-12 hours
  Ascending colon emptying T1/2
Colonic permeability | 2-24 hours after sugars ingestion
  Cumulative excretion of lactulose
Colonic permeability | 8 to 24 hours after ingestion of sugars
  Hourly excretion of mannitol
Small bowel transit time | 6 hours
  Colonic filling at 6 hours (%)
Gastric emptying | 0-2 hours
  Gastric emptying T1/2
Colonic inflammatory response | 4 weeks
  Sigmoid colon mucosal immunocyte count in lamina propria
Stool frequency and consistency | 6 weeks
  Bowel pattern diary
Small bowel inflammatory response | 4 weeks
  Duodenal mucosal immunocyte count in lamina propria

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Vazquez-Roque MI, Camilleri M, Smyrk T, Murray JA, Marietta E, O'Neill J, Carlson P, Lamsam J, Janzow D, Eckert D, Burton D, Zinsmeister AR. A controlled trial of gluten-free diet in patients with irritable bowel syndrome-diarrhea: effects on bowel frequency and intestinal function. Gastroenterology. 2013 May;144(5):903-911.e3. doi: 10.1053/j.gastro.2013.01.049. Epub 2013 Jan 25. PMID 23357715